CLINICAL TRIAL: NCT05873777
Title: 68Ga-FAPI-LM3 PET/CT Imaging in Patients With FAP/SSTR2 Positive Disease and Compared With 18F-FDG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMFHIIT-2022SL070
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: SSTR2; FAP; Positron-Emission Tomography
Keywords: SSTR2; FAP; Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Subjects with malignant diseases (either FAP or SSTR2 positive expression) undergo contemporaneous 68Ga-FAPI-LM3 and 18F-FDG PET/CT for diseases assessment. A part of participants will also undergo additional 68Ga-FAPI-46 PET/CT for comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI-LM3 (Experimental): Each subject receives a single intravenous injection of 18F-FDG and 68Ga-FAPI-LM3, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 18F-FDG PET/CT, 68Ga-FAPI-LM3 PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT, 68Ga-FAPI-LM3 PET/CT — Each subject receives a single intravenous injection of 18F-FDG and 68Ga-FAP-LM3, and undergo PET/CT imaging within the specified time. A part of participants will undergo additional 68Ga-FAPI-46 PET/CT for comparison.

SUMMARY:
As a new dual receptor (SSTR2 and FAP) targeting PET radiotracer, 68Ga-FAPI-LM3 is promising as an excellent imaging agent applicable to SSTR2 positive diseases. In this research, we investigate the safety, biodistribution and radiation dosimetry of 68Ga-FAPI-LM3 in healthy volunteers. Moreover, we evaluate the potential usefulness of 68Ga-FAPI-LM3 positron emission tomography/computed tomography (PET/CT) for the diagnosis of lesions in SSTR2 positive diseases, and compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
As a new dual receptor (SSTR2 and FAP) targeting PET radiotracer, 68Ga-FAPI-LM3 is promising as an excellent imaging agent applicable to SSTR2 positive diseases In this research, we investigate the safety, biodistribution and radiation dosimetry of 68Ga-FAPI-LM3 in healthy volunteers. Moreover, subjects with SSTR2 positive diseases underwent contemporaneous 68Ga-FAPI-LM3 and 18F-FDG PET/CT for diseases assessment. Lesions uptakes were quantified by the maximum standard uptake value (SUVmax). The numbers of positive lesions of 18F-FDG and 68Ga-FAPI-LM3 PET/CT were recorded by visual interpretation. The diagnostic accuracy of 68Ga-FAPI-LM3 were calculated and compared to 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order);
* (ii) patients with suspected or newly diagnosed or previously malignant disease, with either FAP or SSTR2 positive expression (supporting evidence may include MRI, CT, and pathology report etc);
* (iii) patients who had scheduled both 18F-FDG and 68Ga-FAPI-LM3 PET/CT scans;
* (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant disease;
* (ii) patients with pregnancy;
* (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity, and accuracy of 18F-FDG and 68Ga-FAPI-LM3 PET/CT were calculated and compared to evaluate the diagnostic accuracy

SECONDARY OUTCOMES:
SUV | 2 days
  Standardized uptake value (SUV) of 18F-FDG and 68Ga-FAPI-LM3 PET/CT for each positive lesion of subject.
Number of lesions | 2 days
  The numbers of positive lesions of 18F-FDG and 68Ga-FAPI-LM3 PET/CT were recorded by visual interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Director — The First Affiliated Hospital of Xiamen University, Fujian, China
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao L, Pang Y, Fang J, Chen J, Zhou Y, Sun L, Wu H, Guo Z, Lin Q, Chen H. Design, Preclinical Evaluation, and Clinical Translation of 68Ga-FAPI-LM3, a Heterobivalent Molecule for PET Imaging of Nasopharyngeal Carcinoma. J Nucl Med. 2024 Mar 1;65(3):394-401. doi: 10.2967/jnumed.123.266183. PMID 38176714